CLINICAL TRIAL: NCT04450225
Title: Testing the Psychometric Properties of the Italian Version of the Reintegration to Normal Living Index in Complex Patients Discharge From Physical Medicine and Rehabilitation Unit: a Validation Study
Brief Title: The Psychometric Properties of the Italian Version of the Reintegration to Normal Living Index in Complex Patients
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: RNLI_MFR_2020
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-02

CONDITIONS: Complex Patient
Keywords: validation study; social participation; rehabilitation; occupational therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Since the post-acute phase, patients have occupational needs related to social reintegration, that improve the autonomy, social roles in family, at work and in the community.

Unmet needs could lead to a lower level of social reintegration. Healthcare professionals should be able to recognize the level of social reintegration of complex patients discharged from the Physical Medicine Rehabilitation (PRM) unit with the aim to identify those who need intervention aimed at improving social reintegration.

The preliminary Italian version of the RNL index (RNLI) will describe the social reintegration level of the target population, once its psychometric properties will be tested.

DETAILED DESCRIPTION:
The investigators will recruit three groups of participants to test the psychometric properties of the Italian version of the RNLI: complex patients, caregivers and stakeholders.

Phase_1: to test the Content validity. The content validity will be tested on 10 complex patients and 10 stakeholders, who will assess the clarity and relevance of the RNLI items, respectively. In this phase, complex patients are hospitalized in the PMR unit.

From this first phase, the investigators will obtain the preliminary Italian version of the RNLI to test its psychometric properties.

Phase_2: to test the Reliability, Construct validity and Responsiveness. During the hospitalization in the PMR unit, 138 patients and their caregivers will be recruited. During this phase, the investigators will detect the important occupational activities of complex patients enrolled through a semi-structured interview conducted in person.

After discharge, the investigators will contact the patients and their caregivers by telephone at different times (T0, T1 and T2) to test the following psychometric properties through the administration of the Italian version of the RNLI and the Canadian Occupational Performance Measure (COPM). Caregiver will have to answer to the RNLI as a proxy for the patient.

The contact times and the psychometric properties that will be tested are:

T0_ 2 weeks after discharge

* internal consistency
* inter-observer reliability
* convergent construct validity

T1_ 10-14 days after T0

- test-retest reliability

T2_ 6-8 weeks after T0

* discriminant construct validity
* responsiveness

ELIGIBILITY:
For patient:

Inclusion Criteria:

* hospitalized in the PMR unit of AUSL-IRCCS of Reggio Emilia
* Rehabilitation Complexity Scale Extended ≥ 9
* Discharge at home

Exclusion Criteria:

* language barrier
* comorbidities that limit communication and/or collaboration (eg aphasia, dementia, cognitive deficits, severe anxious-depressive syndromes pre-existent to hospitalization, etc.)
* discharge in residential structures, retirement homes or long-term care or transferred to acute wards for complications.

For caregiver:

main caregivers of the patients enrolled

For stakeholders:

a rehabilitation healthcare professional with at least 3 years of clinical experience in rehabilitation and reintegration into the living environment of highly complex patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients admitted to the PMR unit of the AUSL-IRCCS of Reggio Emilia are patients with: disability connected to oncological pathologies, stroke or cerebral hemorrhage outcomes, outcomes of orthopedic interventions for polytrauma or femur fracture, outcomes of brain, spinal or spine neurosurgical operations, limb amputations or acute disabling neurological pathologies (e.g. Guillain-Barrè syndrome, etc.). The length of hospitalization on average is 22.5 days. The percentage of return to home after discharge is 85%, while 9% of patients are discharged to residential structures, retirement homes or long term care. Six percent of patients are transferred back to acute wards for complications.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase_1: to test the Content validity of the Reintegration to Normal Living Index | 3 months
  A group of complex patients and stakeholders will report the clarity and the relevance of the items of the Reintegration to Normal Living Index (RNLI), respectively. Thus, the content validity of the RNLI will be tested.

SECONDARY OUTCOMES:
Phase_2: to test the Reliability, Construct validity and Responsivness of the Reintegration to Normal Living Index | 19 months
  The Reintegration to Normal Living Index (RNLI) and the Canadian Occupational Performance Measure (COPM) will be administer to the complex patients and their caregiver in different times to test the psychometric properties of the RNLI.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Pellegrini, Principal Investigator — AUSL of Reggio Emilia
Locations (1):
- Azienda Unità Sanitaria Locale - IRCCS, Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No